CLINICAL TRIAL: NCT04798755
Title: Efficacy, Safety and Cost-effectiveness of Methotrexate, Adalimumab, or Their Combination in Non-infectious Non-anterior Uveitis: a Randomized, Parallel 3 Arms, Active-controlled, Phase 3 Open Label With Blinded Outcome Assessment Study
Brief Title: Efficacy, Safety and Costs of Methotrexate, Adalimumab, or Their Combination in Non-infectious Non-anterior Uveitis
Acronym: Co-THEIA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Luis Rodriguez Rodriguez, Principal Investigator, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Co-THEIA
Record Dates: First submitted 2021-03-09; First posted 2021-03-15 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis | interventions — Methotrexate; Adalimumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adalimumab (Active Comparator)
  Interventions: Drug: Adalimumab
- Methotrexate (Active Comparator)
  Interventions: Drug: Methotrexate
- Adalimumab+Methotrexate (Experimental)
  Interventions: Drug: Adalimumab+Methotrexate

INTERVENTIONS:
Drug: Methotrexate — Inicial dose 15mg/week increasing up to 25 mg/week
  Arms: Methotrexate
Drug: Adalimumab — At the Baselin visit adalimumab 80 mg subcutaneous loading dose followed a week later by 40 mg every-other-week starting at Week 1.
  Arms: Adalimumab
Drug: Adalimumab+Methotrexate — Adalimumab: at the Baseline visit 80 mg subcutaneous loading dose followed a week later by 40 mg every-other-week starting at Week 1.
  Methotrexate:Inicial dose 15mg/week increasing up to 25 mg/week
  Arms: Adalimumab+Methotrexate

SUMMARY:
Introduction: Non-infectious uveitis (NIUs) include a heterogeneous group of sight-threatening conditions. NIUs can be highly disabling and be associated with a profound impact in the quality-of-life (QoL) and wellbeing. Their correct management sometimes requires the use of immunosuppressive drugs (ISDs), which can be prescribed in monotherapy or in combination. Several observational studies have provided evidence that the use of ISDs in combination could be more effective than and as safe as their use in monotherapy. However, a direct comparison between these two treatment strategies has not been carried out yet.

Methods and analysis: The Combination THerapy with mEthotrexate and adalImumAb for uveitis (CoTHEIA) study is a phase III, multicenter, prospective, randomized, single-blinded with masked outcome assessment, parallel three arms with 1:1:1 allocation, active-controlled, superiority study design, comparing the efficacy, safety and cost-effectiveness of methotrexate (MTX), adalimumab (ADA), or their combination in non-infectious non-anterior uveitis. The duration of the treatment and follow-up will last up to 52 weeks. The complete and maintained resolution of the ocular inflammation will be assessed by masked evaluators (primary outcome). In addition to other secundray measures of efficacy (QoL, visual acuity, costs) and safety, we will identify subjects' subgroups with different treatment responses by developing prediction models based on machine learning techniques using genetic and proteomic biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed with non-infectious intermediate-, posterior-, or pan-uveitis in at least one eye;
2. Adult patients (≥18 years);
3. Subjects with at least one flare of active eye inflammation in the previous 180 days before Baseline visit, defined by the presence of at least 1 of the following parameters in either eye:

   1. Active chorioretinal or retinal vascular lesion, AND/OR
   2. Presence of macular edema by optical coherence tomography (OCT:thickness >350 μm AND cysts or intraretinal fluid), AND/OR
   3. ≥ 2+ anterior chamber cells (ACC; SUN criteria4) , AND/OR
   4. ≥ 2+ vitreous haze (National Eye Institute [NEI]113/SUN criteria4).
4. Subjects with active eye inflammation at Baseline visit, defined by the presence of at least 1 of the following parameters in either eye:

   1. Active chorioretinal or retinal vascular lesion, AND/OR
   2. Presence of macular edema by OCT (thickness >350 μm AND cysts or intraretinal fluid), AND/OR
   3. ≥ 1+ ACC, AND/OR
   4. ≥ 1+ vitreous haze.
5. Subjects meeting at least ONE of the following criteria:

   1. Subjects with known chronic condition necessitating GCs-sparing immunosuppressive treatment: Behçet's disease with posterior segment involvement, multifocal choroiditis with panuveitis, serpiginous choroidopathy, birdshot retinochoroidopathy, diffuse retinal vasculitis, Vogt-Koyanagi-Harada with bullous serous retinal and/or choroidal detachments, sympathetic ophthalmia. No prior therapy is required for these patients. AND/OR
   2. Subjects with registered local/systemic corticosteroid refractory uveitis in the previous 180 months before Baseline visit, defined as:

      * Presence of active inflammation after 4 weeks of high-dose (1mg/kg prednisone equivalent) corticosteroid treatment, resulting in an incomplete response (there was an amelioration, but there is still inflammation); AND/OR, Presence of active inflammation 4 weeks after a regional corticosteroid injection; AND/OR,
      * Treatment with oral corticosteroids resulting in a reduction of inflammation, followed by relapse [increase in ≥1 grade in ACC or vitreous haze or a change of non-active to active lesions (including chorioretinal or retinal vascular lesion and/or macular edema)] when GCs was tapered; AND/OR,
      * Presence of active inflammation after a long-acting corticosteroid intramuscular injection administered between 4 weeks to 180 days before the Baseline visit); AND/OR, Active inflammation after treatment with >10mg/day oral prednisone for at least the past 90 days before Baseline.
6. If female, subject is:

   1. Not of childbearing potential: at least 1 year or more since the final menstrual period or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy);
   2. Of childbearing potential and willing to use an acceptable method of contraception during the study period (i.e. pharmacologics, devices, barrier methods) or abstinence, and for 150 days after the last dose of study drugs;
   3. Not pregnant or breastfeeding
7. Subject has a negative tuberculosis skin test (PPD test or equivalent) and nonpathological Chest X-ray (CXR; Posterior-anterior and lateral view) at Screening or in the previous 90 days before Baseline visit. If the subject has a positive PPD test (or equivalent), has had a past ulcerative reaction to PPD placement and/or a CXR consistent with prior tuberculosis (TB) exposure, the subject must initiate, be currently receiving or have documented completion of a course of prophylactic anti-TB therapy
8. Subjects able and willing to provide written informed consent and to comply with the study protocol.
9. Do not participate in another clinical trial.

Exclusion Criteria:

1. Subjects with confirmed or suspected infectious uveitis, including ocular histoplasmosis syndrome
2. Subjects with previous intolerability, safety issues according to investigator criteria, AND/OR previous failure to control ocular or other inflammation with MTX
3. Subjects with previous exposure to any biological therapy at any time (excluding intravitreal anti-vascular endothelial growth factor [anti-VEGF] therapy and denosumab), including those with that have a potential or known association with progressive multifocal leukoencephalopathy (i.e. natalizumab, rituximab or efalizumab);
4. Subjects with previous exposure to synthetic immunosuppressive therapy (such as mycophenolate or cyclosporine) other than corticosteroids in the past 6 months before Baseline;
5. Subjects with chronic structural eye damage considered by the Site's

Investigator to:

a. Interfere with the measurement of any of the study outcomes, AND/OR b. Cause eye damage regardless of the inflammatory process, AND/OR c. Prevent the normalization of the eye structures; 6. Chronic hypotony (IOP < 5 mm Hg for in the last 3 months and/or in the baseline visit) in both eyes; 7. Subjects receiving local GCs 8. Subjects receiving intravitreal anti-VEGF therapy 9. Subjects with a history of prior intraocular surgery within 30 days prior to the Baseline visit, AND/OR any planned eye surgery within the next 52 weeks from Baseline Visit 10. Subjects with best spectacle-corrected visual acuity (BCVA) worse than 20/400 (ETDRS logMAR > 1.34) in the better eye during the screening or at Baseline visit 11. Subjects with active malignancy considered by the Site's Investigator, including lymphoma, leukemia, non-melanoma skin cancer, and confirmed or suspected ocular masquerade syndromes 12. Subjects with systemic autoimmune disease or ocular condition (besides uveitis) anticipated to dictate treatment course, as considered by the Site's Investigator 14. Subjects with systemic active or chronic recurring infections, such as active TB, syphilis, or hepatitis B or C, at Screening visit or in the previous 90 days before Baseline visit; AND/OR a history of invasive infection (e.g., listeriosisand histoplasmosis); 15. Subjects with history of moderate to severe congestive heart failure (NYHA class III or IV), recent cerebrovascular accident (6 months) and any other condition which, in the opinion of the Site's Investigator, would put the subject at risk by participation in the study 16. Subjects with clinically significant abnormal screening laboratory results as evaluated by the Site's Investigator (at screening/baseline or in the previous4 weeks).

17. Central nervous system demyelinating disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Good Clinical Response | 52 weeks
  Complete resolution of the ocular inflammatory signs, achieved within the first 16 weeks of the study, and maintained until week 52; no treatment failure due to safety or intolerability.

SECONDARY OUTCOMES:
Good Clinical Response | week 16
  Complete resolution of the ocular inflammatory signs, achieved within the first 16 weeks of the study, and maintained until week 52; no treatment failure due to safety or intolerability.
EuroQol-5D at each study visit | Baseline, weeks 16 and 52.
  We will use the EuroQol-5D (0-100, the higher the better quality of life) to compare the change in health-related quality of life between treatment strategies.
Visual Functioning Questionnaire-25 (VFQ-25) | Baseline, weeks 16 and 52.
  We will use the VFQ-25 (0-100, the higher the better quality of life) to compare the change in visual-related quality of life between treatment strategies
Hospital Anxiety and Depression Scale; HADS | Baseline, weeks 16 and 52.
  We will use the HADS (0-21 for either anxiety or depression, the higher the more severe anxiety/depression symptoms) to compare the change in anxiety and depression sympthoms between treatment strategies quality of life, anxiety and depression) between treatment strategies
Clinical components of the Good Clinical Response variable | Baseline, weeks 16 and 52.
  Presence of non active chorioretinal lesions; active retinal vascular inflammation; macular edema; ACC; vitreous haze; and loss of CVA secondary to inflammation
Time to inflammatory relapse. | week 16.
  time from visit 16 weeks until end of the study, loss of follow-up or appearance of at least one ocular inflammatory manifestation, in those individuals achieving a Good Clinical Response.
Best corrected visual acuity (BCVA) | Baseline, weeks 16 and 52.
  We will use the BCVA between treatment strategies
Anti-ADA antibodies (AAA). | Weeks 15, 27 and 51.
  Presence of anti-ADA antibodies (AAA) in subjects receiving this study drug.
Cost-efficacy | Week 52.
  Direct and indirect cost, and Incremental Cost Effectiveness Ratios
Safety: adverse events. | Baseline, weeks 16 and 52.
  Ocurrence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Rodriguez Rodriguez, Principal Investigator — Fundación para la Investigacion Biomédica del Hospital Clínico San Carlos
Locations (14):
- Spain (14):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Cruces, Barakaldo
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria
  - Complejo Asistencial Universitario de León, León
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes
  - Complejo Hospitalario Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Doctor Peset, Valencia
  - Instituto Universitario de Oftalmología Aplicada, Valladolid

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in uveitis. Data or samples shared will be coded, and donated to a Registered Biobank and made available under legal requirement. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
  Regarding dissemination, in order to communicate the clinical trial progress and findings to a broad group of stakeholders, we will elaborate a Dissemination plan which will include production of materials adapted to scientific meetings, scientific publications, patients, and other stakeholders. A summary of the final version of the study protocol will be made available through the Spanish Clinical Trial Registry (REEC) and Clinicaltrials.gov database. The promoter will be the only with access to the participant-level data, following the regulation on data protection.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Derived] Rivas AB, Lopez-Picado A, Calamia V, Carreno E, Cocho L, Cordero-Coma M, Fonollosa A, Francisco Hernandez FM, Garcia-Aparicio A, Garcia-Gonzalez J, Mondejar JJ, Lojo-Oliveira L, Martinez-Costa L, Munoz S, Peiteado D, Pinto JA, Rodriguez-Lozano B, Pato E, Diaz-Valle D, Molina E, Tebar LA, Rodriguez-Rodriguez L; CoTHEIA Study Group. Efficacy, safety and cost-effectiveness of methotrexate, adalimumab or their combination in non-infectious non-anterior uveitis: a protocol for a multicentre, randomised, parallel three arms, active-controlled, phase III open label with blinded outcome assessment study. BMJ Open. 2022 Mar 22;12(3):e051378. doi: 10.1136/bmjopen-2021-051378. PMID 35318229